CLINICAL TRIAL: NCT01576549
Title: An Exploratory Open-Label Biomarker Study of LY2127399 in Patients With Moderate to Severe Rheumatoid Arthritis Receiving Synovial Biopsies
Brief Title: A Study of LY2127399 in Rheumatoid Arthritis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Insufficient efficacy observed in study BCDM(NCT01198002) and BCDV(NCT01202773).
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14319; H9B-MC-BCEE (Other: Eli Lilly and Company)
Record Dates: First submitted 2012-04-10; First posted 2012-04-12 (Estimated); Results first posted 2018-04-26 (Actual); Last update posted 2018-04-26 (Actual); Status verified 2018-03

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tabalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LY2127399 (Experimental): LY2127399 given subcutaneously (SC) at 240 milligrams (mg) as a loading dose in the first week followed by 120 mg SC every 4 weeks for up to 52 weeks.
  Interventions: Drug: LY2127399

INTERVENTIONS:
Drug: LY2127399 — Administered subcutaneously
  Other Names: tabalumab

SUMMARY:
This study will investigate how LY2127399 works in participants with rheumatoid arthritis (RA) who are not adequately responding to methotrexate. Participants will receive LY2127399 via an injection(s) under the skin at 4 week intervals for up to 52 weeks. Key study procedures include biopsies of the lining of an inflamed joint and blood tests to measure RA activity.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of adult onset RA disease according to revised 1987 American Rheumatism Association (ARA) criteria and currently have a documented history of positive for rheumatoid factor (RF) and/or anti-cyclic citrullinated peptide antibody (anti-CCP Ab) and have moderately to severely active RA despite ongoing methotrexate (MTX) therapy
* Have active RA defined as the presence of at least 8/68 tender and at least 8/66 swollen joints, as determined by the tender joint count and swollen joint count assessment forms
* Have a screening C-reactive protein (CRP) measurement greater than 1.2 times upper limit of normal or erythrocyte sedimentation rate (ESR) greater than 28 millimeters/hour (mm/hr)
* Have a clinically inflamed joint suitable for synovial biopsy procedure

Exclusion Criteria:

* Have used an unstable dose of non-steroidal anti-inflammatory drugs (NSAIDs) within 6 weeks prior to baseline
* Have used oral corticosteroids at average daily doses of >10 milligrams/day (mg/day) of prednisone or its equivalent within 6 weeks prior to baseline
* Have received any parenteral corticosteroid injection within 6 weeks of baseline
* Have used other disease-modifying anti-rheumatic drugs (DMARDs) other than MTX, hydroxychloroquine, and/or sulfasalazine in the 8 weeks prior to baseline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2012-05; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (4):
- United States (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Frederick, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Battle Creek, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mayfield, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mesquite, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- LY2127399: Participants received 240 milligrams (mg) LY2127399 administered subcutaneously (SC) (2 SC injections of 120 mg) as a loading dose on Day 1.
  Follow-up visits occurred up to 24 weeks after the final injection of study drug.
Period: Overall Study
Arm/Group | LY2127399
Started | 2
Received at Least 1 Dose of Study Drug | 2
Completed Post-Treatment Follow-Up | 2 (Each participant discontinued dosing and completed the Post-Treatment Follow-Up Period.)
Completed | 0
Not Completed | 2
Not completed — Sponsor Decision | 2

BASELINE CHARACTERISTICS:
Population: Participants who received at least one dose of study drug (LY2127399).
Groups:
- LY2127399: Participants received 240 mg LY2127399 administered SC (2 SC injections of 120 mg) as a loading dose on Day 1.
Arm/Group | LY2127399
Number analyzed (Participants) | 2
Age, Continuous [Mean (Full Range); unit: years] | 66 [52 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Synovitis Scores From Baseline up to Week 16
Description: Primary and secondary analyses were not conducted given insufficient data due to termination of the trial.
Time Frame: Baseline up to Week 16
Population: No participant had outcome measure data analyzed due to the termination of the trial and insufficient sample collection.
Arm/Group | LY2127399
Number analyzed (Participants) | 0

2. Primary Outcome: Percent Change in Synovial B Cell Mass From Baseline up to Week 16
Description: Primary and secondary analyses were not conducted given insufficient data due to termination of the trial.
Time Frame: Baseline up to Week 16
Population: No participant had outcome measure data analyzed due to the termination of the trial and insufficient sample collection.
Arm/Group | LY2127399
Number analyzed (Participants) | 0

3. Primary Outcome: Percent Change in Synovial Immunoglobulin (Ig) Synthesis From Baseline up to Week 16
Description: Primary and secondary analyses were not conducted given insufficient data due to termination of the trial.
Time Frame: Baseline up to Week 16
Population: No participant had outcome measure data analyzed due to the termination of the trial and insufficient sample collection.
Arm/Group | LY2127399
Number analyzed (Participants) | 0

4. Secondary Outcome: Percent Change in Various Cell Types in the Blood From Baseline up to Week 24
Description: Primary and secondary analyses were not conducted given insufficient data due to termination of the trial.
Time Frame: Baseline up to Week 24
Population: No participant had outcome measure data analyzed due to the termination of the trial and insufficient sample collection.
Arm/Group | LY2127399
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Groups:
- LY2127399 - Treatment Period: Participants received 240 mg LY2127399 administered SC (2 SC injections of 120 mg) as a loading dose on Day 1.
- LY2127399 - Follow-up Period: Participants received 240 mg LY2127399 administered SC (2 SC injections of 120 mg) as a loading dose on Day 1.
  Participants then discontinued dosing as a result of study closure, but completed the Post-Treatment Follow-Up Period for up to 24 weeks after the final injection of study drug.
Arm/Group | LY2127399 - Treatment Period | LY2127399 - Follow-up Period
Serious Adverse Events (participants affected / at risk) | 1/2 | 1/2
Other Adverse Events (participants affected / at risk) | 2/2 | 1/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY2127399 - Treatment Period (N=2) | LY2127399 - Follow-up Period (N=2)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY2127399 - Treatment Period (N=2) | LY2127399 - Follow-up Period (N=2)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Rosacea (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Due to early termination of the trial (February 2013 in conjunction with the FLEX RA program), no participant had outcome measure data analyzed. Participants who received study treatment had disposition, demographic, and adverse event data reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days